CLINICAL TRIAL: NCT02836249
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Tenofovir Alafenamide (TAF) 25 mg QD Versus Tenofovir Disoproxil Fumarate (TDF) 300 mg QD for the Treatment of HBeAg Positive, Chronic Hepatitis B
Brief Title: Tenofovir Alafenamide Versus Tenofovir Disoproxil Fumarate for Treatment of Hepatitis B e Antigen-Positive Hepatitis B (China)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-320-0110 (China); 2013-000636-10 (EudraCT Number)
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: HBV; Chronic HBV Infection
Keywords: Hepatitis; Tenofovir; Viread
MeSH Terms: conditions — Hepatitis | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind TAF (Experimental): Tenofovir alafenamide (Vemlidy®; TAF) 25 mg tablet + tenofovir disoproxil fumarate (Viread®; TDF) placebo tablet once daily for up to 144 weeks (per amendment 3.1).
  Interventions: Drug: TAF; Drug: TDF Placebo
- Double-Blind TDF (Active Comparator): TDF 300 mg tablet + TAF placebo tablet once daily for up to 144 weeks (per amendment 3.1).
  Interventions: Drug: TDF; Drug: TAF Placebo
- Open-label TAF (Experimental): All participants who complete the double-blind period will be eligible to receive open-label TAF until Week 384 of the study.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — TAF 25 mg tablet administered orally once daily
  Other Names: GS-7340; Vemlidy®
  Arms: Double-Blind TAF; Open-label TAF
Drug: TDF — TDF 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: Double-Blind TDF
Drug: TAF Placebo — TAF placebo tablet administered orally once daily
  Arms: Double-Blind TDF
Drug: TDF Placebo — TDF placebo tablet administered orally once daily
  Arms: Double-Blind TAF

SUMMARY:
The primary objective of this study is to compare the efficacy, safety, and tolerability of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in treatment-naive and treatment-experienced adults with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B virus (HBV) infection in China.

DETAILED DESCRIPTION:
This study GS-US-320-0110 is an international study planned to enroll participants in global countries, including China. However, due to the review timeline difference in China, full enrollment was reached in the main study (NCT01940471) before China was able to participate. Therefore, this registration only includes the China cohorts as they were not part of the main study analysis. Data for China cohorts were analyzed separately after the main study analysis was completed.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Adult males and non-pregnant, non-lactating females
* Documented evidence of chronic HBV infection
* HBeAg-positive, chronic hepatitis B with all of the following:

  * HBeAg-positive at screening
  * Screening HBV DNA ≥ 2 x 10^4 IU/mL
  * Screening serum alanine aminotransferase (ALT) level > 60 U/L (males) or > 38 U/L (females) and ≤ 10 x the upper limit of the normal range (ULN)
* Treatment-naive participants (defined as < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue) OR treatment-experienced participants (defined as participants meeting all entry criteria [including HBV DNA and serum ALT criteria] and with ≥ 12 weeks of previous treatment with any nucleoside or nucleotide analogue)
* Previous treatment with interferon (pegylated or non-pegylated) must have ended at least 6 months prior to the baseline visit
* Adequate renal function
* Normal ECG

Key Exclusion Criteria:

* Females who are breastfeeding
* Males and females of reproductive potential who are unwilling to use an "effective", protocol specified method(s) of contraception during the study
* Co-infection with hepatitis C virus, HIV, or hepatitis D virus
* Evidence of hepatocellular carcinoma
* Any history of, or current evidence of, clinical hepatic decompensation
* Abnormal hematological and biochemical parameters, including aspartate aminotransferase (AST) > 10 x ULN
* Received solid organ or bone marrow transplant
* History of malignancy within the past 5 years, with the exception of specific cancers that are cured by surgical resection; individuals under evaluation for possible malignancy are not eligible
* Currently receiving therapy with immunomodulators (eg, corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion
* Individuals receiving ongoing therapy with drugs not to be used with tenofovir alafenamide or tenofovir disoproxil fumarate or individuals with a known hypersensitivity to study drugs, metabolites, or formulation excipients
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (25):
- China (25):
  - Beijing Ditan Hospital, Beijing
  - PLA 302 Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Xianya Hospital, Central South University, Changsha
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Nanfang Medical University, Nanfang Hospital, Guangzhou
  - No. 3 Hospital, Zhongshan Medical University, Guangzhou
  - The Affiliated Hospital of Guiyang Medical College, Guiyang
  - The People's Hospital of Hainan Province, Haikou
  - The Second Xiangya Hospital of Central South University, Hunan
  - The First Affiliated Hospital of Nanchang University, Jiangxi
  - 1st Hospital Jilin University, Jilin
  - Jinan Infectious Disease Hospital, Jinan
  - 2nd Hospital of Nanjing City, Nanjing
  - Jiangsu Province People's Hospital, Nanjing
  - Ruijin Hospital, JiaoTong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - 85 Hospital of People's Liberation Army, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Sixth People's Hospital of Shenyang, Shenyang
  - 3rd Hospital of Hebei Medical University, Shijiazhuang
  - West China Hospital, Sichuan University, Sichuan
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - 1st Affiliated Hospital Kunming Medical College, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Hou J, Ning Q, Duan Z, Chen Y, Xie Q, Wang FS, Zhang L, Wu S, Tang H, Li J, Lin F, Yang Y, Gong G, Flaherty JF, Gaggar A, Mo S, Cheng C, Camus G, Chen C, Huang Y, Jia J, Zhang M; GS-US-320-0110 and GS-US-320-0108 China Investigators. 3-year Treatment of Tenofovir Alafenamide vs. Tenofovir Disoproxil Fumarate for Chronic HBV Infection in China. J Clin Transl Hepatol. 2021 Jun 28;9(3):324-334. doi: 10.14218/JCTH.2020.00145. Epub 2021 Apr 28. PMID 34221918
- [Background] Hou J, Ning Q, Duan Z, Chen Y, Xie Q, Zhang L, Wu S, Tang H, Li J, Lin F, Yang Y, Gong G, Luo Y, Xie S, Wang H, Mateo R, Yazdi T, Abramov F, Yee LJ, Flaherty J, Chen C, Huang Y, Zhang M, Jia J. Five-year Treatment with Tenofovir Alafenamide Achieves High Rates of Viral Suppression, Alanine Aminotransferase Normalization, and Favorable Bone and Renal Safety in Chinese Chronic Hepatitis B Patients. J Clin Transl Hepatol. 2024 May 28;12(5):469-480. doi: 10.14218/JCTH.2023.00417. Epub 2024 Apr 15. PMID 38779514
- [Derived] Lim YS, Chan HLY, Ahn SH, Seto WK, Ning Q, Agarwal K, Janssen HLA, Pan CQ, Chuang WL, Izumi N, Fung S, Shalimar, Brunetto M, Hui AJ, Chang TT, Lim SG, Abramov F, Flaherty JF, Wang H, Yee LJ, Kao JH, Gane E, Hou J, Buti M. Tenofovir alafenamide and tenofovir disoproxil fumarate reduce incidence of hepatocellular carcinoma in patients with chronic hepatitis B. JHEP Rep. 2023 Jul 13;5(10):100847. doi: 10.1016/j.jhepr.2023.100847. eCollection 2023 Oct. PMID 37771546
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-320-0110%20(China)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in China.
Pre-assignment Details: 226 participants were screened in China.
Groups:
- Double-Blind: TAF 25 mg: Tenofovir alafenamide (Vemlidy®; TAF) 25 mg tablet + tenofovir disoproxil fumarate (Viread®; TDF) placebo tablet once daily for up to 144 weeks (per amendment 3.1).
- Double-Blind: TDF 300 mg: TDF 300 mg tablet + TAF placebo tablet once daily for up to 144 weeks (per amendment 3.1).
- Open-label: TAF 25 mg to TAF 25 mg: After Week 144 in the Blinded Treatment Phase, participants were given the option to continue with Open-label (OL) TAF 25 mg for additional 240 weeks (Up to Week 384).
- Open-label: TDF 300 mg to TAF 25 mg: After Week 144 in the Blinded Treatment Phase, participants were given the option to switch to OL TAF 25 mg for additional 240 weeks (Up to Week 384).
Period: Double-Blind Treatment Phase
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg | Open-label: TAF 25 mg to TAF 25 mg | Open-label: TDF 300 mg to TAF 25 mg
Started | 123 | 58 | 0 | 0
Completed | 114 | 52 | 0 | 0
Not Completed | 9 | 6 | 0 | 0
Not completed — Randomized but Never Treated | 0 | 1 | 0 | 0
Not completed — Pregnancy | 3 | 1 | 0 | 0
Not completed — Withdrew Consent | 5 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Investigator's discretion | 0 | 1 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0
Period: Open-Label TAF Treatment Phase
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg | Open-label: TAF 25 mg to TAF 25 mg | Open-label: TDF 300 mg to TAF 25 mg
Started (At the end of Double-blind Phase, participants were given the option to receive TAF in an OL TAF Extension Phase for additional 240 weeks.) | 0 | 0 | 113 (Out of 114 participants who completed the Double-blind Phase in TAF 25 mg arm, 1 participant did not enter the OL TAF Extension Phase.) | 52
Completed | 0 | 0 | 100 | 48
Not Completed | 0 | 0 | 13 | 4
Not completed — Lost to Follow-up | 0 | 0 | 6 | 1
Not completed — Withdrew consent | 0 | 0 | 4 | 3
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug. Participants were analyzed according to the treatment they actually received during the double-blinded phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg | Total
Number analyzed (Participants) | 123 | 57 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 121 | 57 | 178
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9.4) | 36 (9.5) | 34 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 48
  Male | 88 | 44 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 123 | 57 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 123 | 57 | 180
HBV DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 7.2 (1.65) | 7.2 (1.48) | 7.2 (1.59)
Plasma HBV DNA Level [Count of Participants; unit: Participants]
  < 8 log10 IU/mL | 74 | 36 | 110
  ≥ 8 log10 IU/mL | 49 | 21 | 70
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 109 | 52 | 161
    CT | 12 | 5 | 17
    TT | 2 | 0 | 2
Oral antiviral (OAV) Treatment Status [Count of Participants; unit: Participants]
  Treatment Experienced | 45 | 18 | 63
  Treatment Naive | 78 | 39 | 117
Proteinuria by Urinalysis (dipstick) [Count of Participants; unit: Participants] — Urine protein was measured using the dipstick method. Grade 0 = Absent; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe
  Participants
    Grade 0 | 117 | 54 | 171
    Grade 1 | 6 | 2 | 8
    Grade 2 | 0 | 1 | 1
    Grade 3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) DNA < 29 IU/mL at Week 48
Time Frame: Week 48
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drugs. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 123 | 57
percentage of participants | 61.0 | 68.4

2. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Seroconversion to Antibody Against Hepatitis B e Antigen (Anti-HBe) at Week 48
Time Frame: Week 48
Population: Serologically Evaluable Full Analysis Set: participants who were randomized, had received at least 1 dose of study drug, and were HBeAg positive and anti-HBe negative or had a value missing value at baseline. Participants were analyzed according to their randomized treatment group. All missing data were treated as no HBeAg seroconversion.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 118 | 57
percentage of participants | 11.0 | 8.8

3. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Hip Dual-Energy X-ray Absorptiometry (DXA) Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline hip BMD values) with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 53 | 31
percent change | 0.624 (2.2731) | -1.507 (2.4193)

4. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline spine BMD values) with available data were analyzed. Dual-energy x ray absorptiometry scans were performed only at sites in China with capability. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 54 | 31
percent change | 0.683 (3.3281) | -2.169 (3.4503)

5. Secondary Outcome: Change From Baseline at Week 48 in Serum Creatinine
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 121 | 55
mg/dL | -0.003 (0.0701) | 0.016 (0.0920)

6. Other Pre Specified Outcome: Percentage of Participants With Treatment-emergent Proteinuria by Urinalysis (Dipstick) Through Week 48
Description: Grades 1 (mild), 2 (moderate), and 3 (severe) were the highest treatment-emergent postbaseline grades for urine protein using the dipstick method.
Time Frame: Up to 48 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg
Number analyzed (Participants) | 123 | 57
percentage of participants
  Grade 1 | 24.4 | 22.8
  Grade 2 | 0.8 | 3.5
  Grade 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to approximately 414 weeks; Adverse Events: Up to Week 384
Description: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug. Participants were analyzed according to the treatment they actually received during the double-blinded phase.
Groups:
- Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg: After Week 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 240 weeks (Up to Week 384).
- Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg: After Week 144 in the Blinded Treatment Phase, participants were given the option to switch to Open-label (OL) TAF 25 mg for additional 240 weeks (Up to Week 384).
Arm/Group | Double-Blind: TAF 25 mg | Double-Blind: TDF 300 mg | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/57 | 1/113 | 0/52
Serious Adverse Events (participants affected / at risk) | 8/123 | 3/57 | 7/113 | 4/52
Other Adverse Events (participants affected / at risk) | 85/123 | 43/57 | 84/113 | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: TAF 25 mg (N=123) | Double-Blind: TDF 300 mg (N=57) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=113) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=52)
Cardiac polyp (Cardiac disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: TAF 25 mg (N=123) | Double-Blind: TDF 300 mg (N=57) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=113) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=52)
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 9 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 2 | 2 | 8 | 3
Hepatic cyst (Hepatobiliary disorders) | 5 | 1 | 0 | 4
Hepatic steatosis (Hepatobiliary disorders) | 10 | 3 | 24 | 18
Covid-19 (Infections and infestations) | 0 | 0 | 45 | 12
Nasopharyngitis (Infections and infestations) | 40 | 12 | 11 | 6
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1 | 4
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 27 | 16 | 20 | 12
Urinary tract infection (Infections and infestations) | 8 | 8 | 2 | 2
Amylase increased (Investigations) | 1 | 3 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1 | 3
Blood parathyroid hormone increased (Investigations) | 5 | 4 | 3 | 1
Creatinine renal clearance decreased (Investigations) | 3 | 3 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 0 | 10 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 2 | 1 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 6 | 5
Dizziness (Nervous system disorders) | 6 | 4 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 4 | 3
Proteinuria (Renal and urinary disorders) | 0 | 4 | 1 | 1
Renal cyst (Renal and urinary disorders) | 2 | 0 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 1
Hypertension (Vascular disorders) | 3 | 1 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT02836249/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT02836249/SAP_001.pdf